CLINICAL TRIAL: NCT06979466
Title: Facilitation Recovery For Patients With Chronic Stroke: The Q Therapeutic System, Frequency-Tuned Electromagnetic Field Treatment
Brief Title: Q Therapeutic System for Chronic Stroke Recovery
Acronym: EMAGINE-C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burke Rehabilitation Hospital (Other)
Collaborators: BrainQ Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRH_EMAGINE C IIT_202501
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Hemorrhage; Brain Injury; Cerebrovascular Accident (CVA); Chronic Stroke Patient
Keywords: BrainQ; Stroke; Cerebrovascular Disorders; Electromagnetic Stimulation
MeSH Terms: conditions — Stroke; Hemorrhage; Brain Injuries; Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, open-label, single center clinical trial designed to evaluate the efficacy, and safety of the intervention in the management of chronic stroke patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BQ 3.0 Active Stimulation Group (Experimental): 60 sessions over a period of 12 weeks (5 treatments per week) of active study intervention with the BQ 3.0 (frequency and intensity parameters will be set to 1-100 Hz.; 0.1-1.0 G), including a standardized, pre-defined and evidence-based physical and occupational therapy regimen concurrent with the study intervention.
  Interventions: Device: Q Therapeutic System (BQ 3.0) - Active

INTERVENTIONS:
Device: Q Therapeutic System (BQ 3.0) - Active — The BQ 3.0 is a medical device that produces and delivers non-invasive, extremely low intensity and frequency (1-100 Hz.; 0.1-1.0 G), frequency tuned electromagnetic fields in order to stimulate neuronal networks with the aim of reducing disability and promoting neurorecovery
  Other Names: BQ 3.0 Active Stimulation Group Interventions

SUMMARY:
Evaluate the effectiveness of the Q Therapeutic (BQ 3.0) System for individuals with chronic stroke in improving upper extremity function as determined by change in functional outcome measures after 3-month treatment, including in-clinic and at-home sessions.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label, single center clinical trial designed to evaluate the safety, feasibility, and efficacy of the Q Therapeutic (BQ 3.0) System in the management of chronic stroke patients. Primarily, the trial will assess the System's impact on the upper extremity function through objective, validated clinical assessments. Secondary endpoints will evaluate additional functional and global disability, quality-of-life and safety outcomes.

The study intervention will consist of a total of 5 sessions per week over a period of 3 months (12 weeks) for a total of up to 60 sessions. Each participant must complete at least 40 sessions over the 12-week period to complete the protocol. No extra time will be given to complete all 60 sessions. Each session will last up to 60 minutes during which 40 minutes of active stimulation using the BQ 3.0 System will be administered to participants. The 40 minutes of stimulation will be paired with seated upper extremity (UE) exercises. Lastly, the device will be removed and 10 minutes of standing balance and LE strengthening exercises will be performed without stimulation. A battery of clinical assessments will be conducted before and after the 60 exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

* FMA-UE score between 22-50 (inclusive) of impaired limb.
* Difference between Screening and Baseline visit FMA-UE is 3 points or fewer.
* Age 18 to 80 years of age (inclusive).
* Stroke due to ischemia or to intracerebral hemorrhage.
* >6 months to 5 years from index stroke onset.
* Box & Block Test score with affected arm is ≥1 block in 60 seconds at Baseline Visit.
* Able to sit with the investigational System for 40 consecutive minutes.
* Can follow a 3-step command, such as "take the paper, fold it in half, and return it to me", or a non-verbal equivalent.
* Willingness to participate in physical exercises during study intervention sessions.
* Availability of a relative or other caregiver able to assist during study treatment sessions and visits.
* If female, not pregnant or breastfeeding or planning pregnancy during the study period.
* Informed consent signed by subject.

Exclusion Criteria:

* Severe neglect impairment interfering with assessments or treatments.
* Severe depression, defined as GDS Score >10/15
* The presence of MR-incompatible implanted devices or MR-incompatible retained objects; or the presence of life-sustaining MR-compatible devices (e.g. pacemaker or internal cardiac defibrillator).
* Active epilepsy or currently taking anti-epileptic medication (indicated for the treatment of a seizure disorder), or any epileptic seizure in the last 5 years
* Botulinum toxin to the paretic arm: received in the prior 3 months OR expected before the 6-Month Visit
* Severe UE spasticity, defined as presence of upper extremity contracture or modified Ashworth Scale score≥3 in either biceps or pectoralis
* Pre-existing neurological condition (eg, Alzheimer's disease, Parkinson's disease, multiple sclerosis, traumatic brain injury, spinal cord injury) or physical limitation that would interfere significantly with the subject's participation in the study and/or confound neurological or functional evaluation.
* Significant visual disturbances, pre-existing or resulting from the index stroke, that cannot be corrected and that would interfere significantly with the subject's participation in the study and/or confound neurological or functional evaluation.
* Unstable serious illness/condition (eg, active cancer, severe heart failure, active major psychiatric condition) or life expectancy of less than 12 months.
* Alcohol abuse and/or illicit drug abuse in the past 6 months, which is likely to influence ability to fully participate in the trial.
* Participation in another interventional trial that would conflict with the current study or clinical endpoint interference may occur.
* Participation in an upper extremity rehabilitation program provided by a licensed provider in the 4 weeks prior to the Screening visit, or a or planned participation in such program at any time between the Screening Visit and the primary endpoint visit.
* Employee of the Sponsor.
* Prisoner.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity | Baseline, 3 month, 5 month, 6 month
  a standardized, performance-based measure used to assess motor impairment in the upper limb following stroke or other neurological injuries

SECONDARY OUTCOMES:
Box and Block Test | Baseline, 3 month, 5 month, 6 month
  Timed test used to assess unilateral gross manual dexterity
Geriatric Depression Scale (Short Form) (GDS) | Baseline, 3 month, 5 month, 6 month
  15-question self-administered questionnaire used to screen for depression in older adults. Each item is answered "Yes" or "No." One point is given for each answer that indicates depression (specific answers are predetermined). Score Range from 0-15. Interpretation: 0-4: Normal (no depression), 5-8: Mild depression, 9-11: Moderate Depression, 12-15: Severe Depression.
modified Rankin Scale (mRS) | Baseline, 3 month, 5 month, 6 month
  Tool to assess the degree of disability or dependence in daily activities following a stroke or other neurological event. Scores range from 0 (no symptoms), 1 (no significant disability) to 6 (death), with increasing scores indicating greater levels of disability.
Stroke Impact Scale (SIS) Hand Domain | Baseline, 3 month, 5 month, 6 month
  Assesses hand function through a self-report questionnaire with specific items focusing on how stroke has affected the individual's ability to use their hands in daily tasks. Each of the five items is rated on a 5-point scale from 1 (could not do at all) to 5 (not difficult at all), transformed to a 0-100 scale, where higher scores indicate better hand function. 0-19 (very severe difficulty or complete inability to use the hand), 20-39 (severe difficulty), 40-59 (moderate difficulty), 60-79 (mild difficulty), 80-100 (minimal or no difficulty with hand function).
Stroke Impact Scale 16 (SIS-16) | Baseline, 3 month, 5 month, 6 month
  16-item instrument designed to assess physical function in individuals with stroke. Each item is rated on a 5-point scale from 1 (could not do it at all) to 5 (not difficult at all) and the total raw score is transformed to a 0-100 scale, with higher scores indicating better physical functioning. 0-19 (very severe limitations, unable to perform most physical tasks independently), 20-39 (severe physical limitations, significant dependence on others), 40-59 (moderate physical limitations, difficult with many daily activities), 60-79 (mild physical limitations, may need some assistance or accommodations), 80-100 (minimal to no physical limitations, high level of independence)
Nine Hole Peg Test (9HPT) | Baseline, 3 month, 5 month, 6 month
  Standardized, quantitative assessment used to evaluate finger dexterity
10 Meter Walk Test (10MWT) | Baseline, 3 month, 5 month, 6 month
  Standardized assessment used to measure gait speed, a key indicator of functional mobility
Functional Ambulation Categories (FAC) | Baseline, 3 month, 5 month, 6 month
  6-point functional walking test that evaluates ambulation ability, determining how much human support the patient requires when walking. Scores range from 0 (non-functional ambulation) to 5 (independent ambulation on all surfaces including stairs). Higher scores indicate greater walking independence
5-level EQ-5D (EQ-5D-5L) | Baseline, 3 month, 5 month, 6 month
  Brief, multi-attribute, generic health status measure that uses a descriptive system and a visual analogue scale (EQ-VAS). Five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is rated on a 5-level scale, from no problems (1) to extreme problems (5), generating a 5-digit health state that is converted into an index value (typically 0 = death to 1 = full health, with possible negative values for health states worse than death). A higher index score indicates better perceived overall health status, and a visual analog scale (VAS) is also included to rate health from 0 (worst) to 100 (best imaginable health).
Berg Balance Scale (BBS) | Baseline, 3 month, 5 month, 6 month
  Non mandatory assessment - 14-item functional test designed to assess balance and risk of falls in older adults, but it can also be used with other populations. Each item is scored from 0 to 4, with a maximum total score of 56, where higher scores indicate better balance. Scores 41-56 suggest low fall risk, 21-40 indicate moderate risk, and 0-20 reflect a high risk of falling and significant balance impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Burke Rehabilitation Hospital, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with the study sponsor.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be shared from July 2025 to Dec 2026 between the site and study sponsor.
Access Criteria: De-identified data in excel spreadsheets will me made available to the study sponsor.

REFERENCES:
- [Background] Weisinger B, Pandey DP, Saver JL, Hochberg A, Bitton A, Doniger GM, Lifshitz A, Vardi O, Shohami E, Segal Y, Reznik Balter S, Djemal Kay Y, Alter A, Prasad A, Bornstein NM. Frequency-tuned electromagnetic field therapy improves post-stroke motor function: A pilot randomized controlled trial. Front Neurol. 2022 Nov 14;13:1004677. doi: 10.3389/fneur.2022.1004677. eCollection 2022. PMID 36452175
- [Background] Saver JL, Duncan PW, Stein J, Cramer SC, Eng JJ, Lifshitz A, Hochberg A, Bornstein NM. EMAGINE-Study protocol of a randomized controlled trial for determining the efficacy of a frequency tuned electromagnetic field treatment in facilitating recovery within the subacute phase following ischemic stroke. Front Neurol. 2023 May 5;14:1148074. doi: 10.3389/fneur.2023.1148074. eCollection 2023. PMID 37213907
- [Background] Segal Y, Segal L, Blumenfeld-Katzir T, Sasson E, Poliansky V, Loeb E, Levy A, Alter A, Bregman N. The Effect of Electromagnetic Field Treatment on Recovery from Ischemic Stroke in a Rat Stroke Model: Clinical, Imaging, and Pathological Findings. Stroke Res Treat. 2016;2016:6941946. doi: 10.1155/2016/6941946. Epub 2016 Feb 1. PMID 26949561
- [Background] Okabe N, Hovanesyan M, Azarapetian S, Dai W, Weisinger B, Parabucki A, Balter SR, Shohami E, Segal Y, Carmichael ST. Theta Frequency Electromagnetic Stimulation Enhances Functional Recovery After Stroke. Transl Stroke Res. 2025 Apr;16(2):194-206. doi: 10.1007/s12975-023-01202-z. Epub 2023 Nov 14. PMID 37962771